CLINICAL TRIAL: NCT00580931
Title: Efficacy of Nicotinamide for the Treatment of Alzheimer's Disease
Brief Title: Safety Study of Nicotinamide to Treat Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Steven Schreiber, Professor of Neurology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIRG-07-61197
Record Dates: First submitted 2007-12-24; First posted 2007-12-27 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: nutraceutical, dementia, cognition, HDAC inhibitor
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects will receive experimental drug in a blinded fashion.
  Interventions: Drug: Nicotinamide
- 2 (Placebo Comparator): Identical in size, shape and color to experimental drug.
  Interventions: Drug: Enduramide placebo

INTERVENTIONS:
Drug: Nicotinamide — 1500 mg twice a day for 6 months
  Other Names: Enduramide
  Arms: 1
Drug: Enduramide placebo — 1 tab twice a day
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether nicotinamide, or vitamin B3, is safe and effective in the treatment of Alzheimer's disease.

DETAILED DESCRIPTION:
The goal of this proposal is to show that, nicotinamide (NA), a B3 vitamin, is safe and effective for the treatment of patients with mild to moderate Alzheimer's disease (AD). NA is known to block the ability of certain proteins to regulate other proteins by removing their acetyl groups. Recent evidence has demonstrated that inhibitors such as NA prevent nerve cell degeneration in models of Huntington's disease (HD), Parkinson's disease and Lou Gehrig's disease (or ALS). Despite these beneficial effects in many different animal models, there have been no studies to date using these inhibitors in AD. In some of our recent studies we found that the potent inhibitor, NA, significantly improves learning and memory in transgenic mice that develop AD. NA treatment also resulted in striking changes in tau, a protein that abnormally accumulates in AD. NA has been extensively used in clinical studies over the last 40 years and is generally safe and well-tolerated. As NA is a safe and readily available vitamin supplement, our recent results provide a strong argument for a study of NA in patients with AD. We therefore propose to treat 50 patients with mild to moderate AD with either NA (1500 milligrams twice a day) or an identical but inactive drug (placebo) for 24 weeks. At 6 week intervals we will assess functions such as learning and memory, and ability to carry out daily activities as well as caregiver reports using standardized tests. We will also perform spinal taps at the beginning and end of the study to measure the level of abnormal tau protein in the cerebrospinal fluid. Blood tests will periodically be done to assess liver function and complete blood counts. The results of this study may provide the basis for a more extensive study of NA for the treatment of mild to moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to DSM-IV criteria
* Mild to moderate dementia based on Mini-Mental State Examination [MMSE] score between 13-25
* Minimum age 50 years
* Brain imaging (computed tomographic scan or magnetic resonance image) within 12 months consistent with a diagnosis of probable AD
* Hachinski Ischemic Score of <4.
* Stable doses of concomitant medications, including cholinesterase inhibitors (ChEIs) and/or memantine.

Exclusion Criteria:

* Dementia due to another cause
* Other neurological or psychiatric diseases
* Pseudodementia
* Unstable medical condition
* Initial treatment within 30 days of screening with a ChEI, memantine or any investigational drug
* History of alcoholism, drug abuse, liver disease, peptic ulcer disease
* Pregnancy, or the potential to become pregnant.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive Subscale | Baseline, 6 wk, 12 wk, 18 wk, 24 wk

CONTACTS AND LOCATIONS:
Overall Officials: Steven S Schreiber, MD, Principal Investigator — Regents of the University of California
Locations (1):
- UC Irvine School of Medicine, Irvine, California, United States